CLINICAL TRIAL: NCT06193733
Title: Dendritic Cell Vaccination to Prevent Hepatocellular Carcinoma Recurrence After Liver Resection-phase II Clinical Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wei-Chen Lee, Principal Investigator, Clinical Professor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202200329A0
Record Dates: First submitted 2023-12-18; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Procedure: injection of the cell therapy product (Experimental): Procedures per cycle (total of 3 cycles):
  8 days before autologous cell injection: Cytapheresis - Autologous cell injection - 2 days after cell injection: lab assessment.
  Interventions: Biological: Autologous Dendritic Cell

INTERVENTIONS:
Biological: Autologous Dendritic Cell — Biological: Immunotherapy with dendritic cells

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common primary liver tumors. Surgical resection remains the first choice of early stage HCC because the result is superior to other treatments and not limited to liver donation. However, liver resection is criticized that tumor recurrent rate is more than 50% in 5 years although the tumors are completely resected. In our large scale study including 1639 patients with liver resection for HCC, the 1-, 3-, and 5-year disease survival were 73.7%, 58.3% and 53.3%, respectively. Currently there are no effective treatment used as adjuvant therapy to prevent HCC recurrence. Dendritic cells (DC) are the most potent professional antigen-presenting cells, and can capture tumor antigens to provoke antigen-specific cytotoxic T-cells. DC pulsed by tumor associated antigens can be used to proceed tumor-specific immunotherapy. Thereafter, DC pulsed HCC tumor-antigens may be used as an adjuvant therapy to prevent HCC recurrence.

ELIGIBILITY:
Inclusion Criteria:

* The patients have curative liver resection for primary or recurrent HCCs which are diagnosed by pathological figures, and the risk nomogram scores of tumor recurrence are ≥ 101 [Hepatitis, score 57; platelet < 100x103 , score72 ; multiple tumors, score 69 ; cirrhosis, score 62 ; microvascular invasion, score 100 ; total tumor volume > 43.3cm3 ,score 90]
* Age ≧20 years old and sign informed consent.
* BCLC stage A-C
* Child-Pugh sore ≤ 6
* Percentage of lymphocytes in peripheral blood ≧12%.
* Performance status ECOG ≦2
* AST and ALT ≦ 5x upper limit of normal.
* Platelet ≥ 80000/mm3
* WBC ≥ 3000/uL
* RBC ≥ 2.5x106/uL
* eGFR ≥ 30ml/min/1.73m2
* The patients must be disease-free after liver resection, which is confirmed by dynamic CT or MRI within 14 days.
* The participates must have early stage or intermediate stage of HCC and receive liver resections to remove the tumors completely.
* The participates must agree to harvest and preserve tumor specimens during operation.

Exclusion Criteria:

* Subjected having other malignancy except HCC are excluded.
* Uncontrolled or clinical significant cardiac diseases.
* Positive for HIV.
* Active bacterial of fungal infections.
* Prior chemotherapy within one month.
* Use of other investigational drug within one month.
* Subjects with systemic steroid treatment within 14 days.
* Subjects in the status of immune deficiency.
* Subjects in the status of autoimmune diseases.
* Subjects with Long-term use of immunosuppressive agents.
* Subjects with checkpoint inhibitor immunotherapy within one month.
* Subjects with local reginal therapy within one month.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-02-19 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | From date of randomization untill the date of radiographic tumor assessment confirm tumor recurrence, assessed up to 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years